CLINICAL TRIAL: NCT02144649
Title: A Comparison of Tangerine and Red Tomato Juice in Men With Prostate Cancer: A Pilot Study
Brief Title: Tangerine or Red Tomato Juice in Treating Patients With Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Riverside Methodist Hospital (Other)
Responsible Party: Principal Investigator, Steven Clinton, Professor of Internal Medicine, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-13166; NCI-2014-01002 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
Keywords: Prostate Cancer; Tangerine Juice; Tomato Juice
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (control, no juice) (No Intervention): Patients consume no tomato juice.
- Group II (tangerine tomato juice) (Experimental): Patients will consume two 5.5 oz. cans of tangerine tomato juice every day until their scheduled surgery. (approximately 4 weeks)
  Interventions: Dietary Supplement: dietary intervention (tangerine tomato juice); Other: questionnaire administration; Other: Correlative studies
- Group III (red tomato juice) (Experimental): Patients consume two cans of red tomato juice daily until their scheduled surgery (approximately 4 weeks).
  Interventions: Dietary Supplement: dietary intervention (red tomato juice); Other: questionnaire administration; Other: Correlative studies

INTERVENTIONS:
Dietary Supplement: dietary intervention (tangerine tomato juice) — Group II will consume two 5.5 oz. cans of tangerine tomato juice every day until their scheduled surgery. (approximately 4 weeks).
  Other Names: Dietary Modification; intervention, dietary
  Arms: Group II (tangerine tomato juice)
Dietary Supplement: dietary intervention (red tomato juice) — Group III will consume two 5.5 oz. cans of red tomato juice every day until their scheduled surgery (approximately 4 weeks).red tomato juice
  Other Names: Dietary Modification; intervention, dietary
  Arms: Group III (red tomato juice)
Other: questionnaire administration — Men enrolled in the study will be asked to complete a 3-Day Food Record and a series of additional questionnaires (urologic symptom and quality of life questionnaire) at home.
  Other Names: Ancillary studiesAll
  Arms: Group II (tangerine tomato juice); Group III (red tomato juice)
Other: Correlative studies — Blood and urine samples at enrollment and blood, urine, and prostate tissue at the time of surgery to determine compliance with the intervention product and tomato phytochemical biodistribution. Additionally, we will correlate each type of tomato juice with lycopene presence in plasma, urine, and tissue provided by subjects on the day of surgery.
  Other Names: laboratory biomarker analysis
  Arms: Group II (tangerine tomato juice); Group III (red tomato juice)

SUMMARY:
This randomized pilot clinical trial compares tangerine and red tomato juice in treating patients with prostate cancer undergoing surgery. A diet high in lycopene, a substance found in tomatoes, may help prevent normal cells from transforming into cancer cells in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a randomized, three-arm pilot clinical trial to determine compliance and safety of daily consumption of tangerine tomato juice or red tomato juice.

SECONDARY OBJECTIVES:

I. To quantify total carotenoids, total lycopene (LYC), cis-LYC, trans-LYC, phytoene, phytofluene, and lycopene metabolites in plasma and prostate tissue in the three groups of men.

II. To evaluate serum biomarkers related to prostate carcinogenesis, including those previously impacted by tomato phytochemicals (testosterone, sex hormone-binding protein [SHBP], insulin-like growth factor [IGF]-I, IGF-binding protein [BP]3, vascular endothelial growth factor [VEGF], and a panel of anti-inflammatory cytokines) by validated assays.

III. To evaluate molecular signatures using the 200 gene quantitative Nano-string nCounter code set (selected genes known to be impacted by dietary components, genes impacted by common prostate genetic and epigenetic damage, and those regulated by testosterone) and micro-ribonucleic acid (RNA) nCounter code set.

IV. To plot the distribution of carotenoid metabolites across the matrix versus the epithelium and cancer versus non-cancer areas of the prostate using matrix-assisted laser desorption ionization (MALDI) imaging of a limited number of samples.

OUTLINE: Patients are randomized to 1 of 3 treatment groups.

GROUP I: Patients consume no tomato juice.

GROUP II: Patients consume two cans of tangerine tomato juice daily until their scheduled surgery (approximately 4 weeks).

GROUP III: Patients consume two cans of red tomato juice daily until their scheduled surgery (approximately 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Have biopsy proven carcinoma of the prostate
* Have chosen a radical prostatectomy for treatment of their disease after the medical team has presented all possible treatment options
* Not be receiving neoadjuvant hormonal or chemotherapy (other clinical trials)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Not currently be taking tomato carotenoid dietary supplements or "alternative" products (e.g., lycopene supplements, Lyc-O-Mato, saw palmetto); vitamin A and beta-carotene supplements are allowed
* Not be allergic to tomatoes or tomato products
* Have plasma total cholesterol < 200 mg/dL
* Plasma triglycerides < 200 mg/dL
* Have blood urea nitrogen and serum creatinine (BUN/Cr) without clinically significant abnormalities after review by the study physicians
* Liver enzymes without clinically significant abnormalities after review by the study physicians
* Complete blood count (CBC) without clinically significant abnormalities after review by the study physicians
* Prothrombin time (PT) without clinically significant abnormalities after review by the study physicians
* Partial thromboplastin time (PTT) without clinically significant abnormalities after review by the study physicians
* International normalized ratio (INR) without clinically significant abnormalities after review by the study physicians
* Voluntarily agree to participate and sign an informed consent document
* Agree to have prostate biopsy blocks provided to the study for evaluation
* Agree to consume a standardized vitamin and mineral supplement and avoid other nutrition, dietary, or alternative medications/supplements for the duration of the study
* Agree to follow a low lycopene and phytoene diet

Exclusion Criteria:

* Have an active malignancy other than prostate cancer that requires therapy
* Have a prostate biopsy with less than 5% cancer involvement
* Have a history of traumatic or surgical castration
* Have plasma total cholesterol > 200 mg/dL
* Have plasma triglycerides > 200 mg/dL
* Have a history of uncontrolled pituitary hormone diseases that currently require varying doses of supplemental hormonal administration (thyroid hormones, adrenocorticotropic hormone [ACTH], growth hormone) or other endocrine disorders requiring varying doses of hormone administration with the exception of diabetes and osteoporosis
* Are planning to start certain medications after the trial enrollment; no new finasteride (Proscar) or other hormonal agents for chemoprevention/treatment of benign prostate hyperplasia (BPH); utilizing new prescription medications for urinary outlet obstructive symptoms will result in discontinuing participation in this study; the use of new non-prescription substances to improve urinary tract symptoms will also result in discontinuing participation (i.e. saw palmetto, other herbal, alternative products); men who are currently taking finasteride or medications (meds) for urinary outlet obstructive symptoms may enroll in the study as long as there is no plan to change the dose in the weeks prior to surgery
* Have a known allergy to tomatoes or have never consumed tomatoes
* Have active metabolic or digestive illnesses such as malabsorptive disorders (Crohn's, Celiac disease, irritable bowel syndrome [IBS]), renal insufficiency, hepatic insufficiency, cachexia, or short bowel syndrome
* Have significant loss of gastrointestinal organs, except for appendix, due to surgery
* Have altered immunity such as autoimmune disorders, clinically significant anemia, hemophilia, and blood dyscrasias

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09-22 (Actual); Study Completion 2016-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity | Up to time of surgery
Compliance of daily consumption of tangerine tomato juice or red tomato juice | Up to time of surgery
Differences in carotenoid levels of biological samples between groups | Up to time of surgery
  Linear regression analysis will be used to examine differences in carotenoid levels of biological samples between groups.

SECONDARY OUTCOMES:
Change in histopathologic markers between the treatment groups | Baseline to time of surgery
  Compared via 3 way analysis of variance (ANOVA) with pairwise comparisons or nonparametric Kruskal-Wallis tests where appropriate.
Change in immunohistochemical markers between the treatment groups | Baseline to time of surgery
  Compared via 3 way ANOVA with pairwise comparisons, or nonparametric Kruskal-Wallis tests where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schwartz, Ph.D., Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - OhioHealth Dublin Methodist Hospital, Dublin, Ohio

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu